CLINICAL TRIAL: NCT00200291
Title: Changes in Food Reinforcement During Obesity Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 3U01DK067861-02S1 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2007-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): Behavioral: hypocaloric low-fat diet
  Interventions: Behavioral: hypocaloric, low-fat diet
- 2 (Placebo Comparator): Behavioral: hypocaloric, low-fat diet
  Interventions: Behavioral: hypocaloric, low-fat diet

INTERVENTIONS:
Behavioral: hypocaloric, low-fat diet — hypocaloric, low-fat diet

SUMMARY:
The reinforcing value of food, or how much a person "wants" a food, is an important determinant of food intake. Thus far, food reinforcement has only been studied in laboratory settings, and no studies have examined whether the reinforcing value of food is altered when dietary changes are made. The chronic deprivation that occurs when a low-calorie, low-fat diet is implemented for weight loss may increase the reinforcing value of all foods, but particularly for restricted high-fat foods. Greater increases in the reinforcing value of high-fat foods relative to low-fat foods may be detrimental for sustaining newly adopted eating behaviors that produce weight loss, whereas greater increases in the reinforcing value of low-fat foods relative to high-fat foods may aid in maintaining healthy eating behaviors. The aim of this application is to measure food reinforcement in a clinical setting to determine if food reinforcement changes when a traditional weight loss diet is prescribed. For this ancillary study, 147 volunteers will be recruited from the 165 overweight and obese women participating in the Program to Reduce Incontinence by Diet and Exercise (PRIDE) at The Miriam Hospital. As part of PRIDE, these participants will be randomized in a 2-to-1 ratio to either a 6-month weight loss intervention or usual care. Assessments of food reinforcement, dietary intake, and weight will occur at 0 and 6 months. Given that the intervention group changes their diet relative to the usual care group, it is hypothesized: 1) the intervention group will have greater increases in the reinforcing value of both high- and low-fat foods than the usual care group from 0 to 6 months; and 2) within the intervention group, decreases in frequency of consumption of high-fat foods will be related to increases in the reinforcing value of high-fat foods from 0 to 6 months. These results will lead to a novel line of research, examining the relationship between food reinforcement and weight loss maintenance, so that diets can be designed to promote changes in food reinforcement that aid in sustaining dietary changes and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Participants from main parent study - PRIDE

Exclusion Criteria:

* Allergic to foods in investigation

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Reinforcing value of low- and high-fat food | 6 months

SECONDARY OUTCOMES:
diet changes and weight loss | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, Principal Investigator — University of Tennessee
Locations (1):
- The Weight Control and Diabetes Research Center, Providence, Rhode Island, United States